CLINICAL TRIAL: NCT03077087
Title: Single-Stage Integra Reconstruction in Burns
Acronym: Integra
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to feasibility issues with completing the study procedure.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A16-734
Record Dates: First submitted 2017-02-27; First posted 2017-03-10 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2019-09

CONDITIONS: Thermal Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-stage Integra (Experimental): Composed of a porous collagen-chondroitin 6-sulfate fibrillary mat covered with a thin sheet of silastic, it serves to cover wound beds of freshly excised burns and allow for the infiltration of fibroblasts, capillaries, and macrophages, essentially creating a "neodermis" while also acting as a barrier against infection and a blockade against heat and moisture loss
  Interventions: Device: thin Integra® (125 cm2)

INTERVENTIONS:
Device: thin Integra® (125 cm2) — 125 cm2 represents approximately 0.7% of an average sized patient's total body surface area. The remaining injury areas would be covered with standard-thickness Integra® only. The donor graft, a 4 cm x 10 cm sheet of skin, would be meshed in a 3:1 ratio to be expanded to cover the 125 cm2 sheet of thin Integra®. The patient's post-operative care would be largely unchanged, although the patient would have a donor site of 40 cm2 that would be dressed and managed in the usual fashion.
  Other Names: Integra®

SUMMARY:
This is a prospective, descriptive, pilot case series involving patients with significant burns who are candidates for reconstruction with Integra®. Subjects would have a small area of the wound would, at the time of excision, have the smallest sheet of thin Integra® (125 cm2) placed and be immediately autografted with a 3:1 meshed split-thickness skin graft. Of note, 125 cm2 represents approximately 0.7% of an average sized patient's total body surface area, so for even the smallest burns in our proposed trial, this area would represent a small portion of the patient's area of injury. The remaining injury areas would be covered with standard-thickness Integra® only.

DETAILED DESCRIPTION:
Integra®, a synthetic dermal substitute, has been utilized in burn care for decades. Typically, 10-14 days after Integra® placement, a patient returns to the operating room, the top silastic layer of the Integra® is removed, and an autograft - a split-thickness skin graft harvested from the patient - is applied directly on top of the incorporated Integra®. The result is regarded to be a cosmetically and functionally superior result to that which would have been obtained had the wound bed itself been autografted at the time of excision, as opposed to being covered by Integra® and autografted during a second operation.

Integra® use in single-stage procedures to cover defects without grafting has shown benefit when defects are fairly small, e.g. fingertip injuries, and small head and neck skin cancer resections. While single-stage reconstruction with Integra® has been demonstrated with standard thickness Integra®, this decreased thickness would increase the likelihood of graft survival due to the decreased distance of nutrient diffusion.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult burn patients greater than 18 years old, admitted with burn injuries eligible for Integra® reconstruction at the discretion of the burn attending physicians.

Exclusion Criteria:

* patients with isolated hand or face burns - these burns are treated with sheet grafts (unmeshed); the 3:1 mesh grafts would not be used on these cosmetically sensitive areas. If they have hand and/or face burns in addition to other areas, they will not be excluded. However, the study itself will not be performed on the hands or face. Additionally, patients unable to present to our clinic for routine follow-up due to geographic limitations or otherwise will be ineligible.

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Mohr, MD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD

REFERENCES:
- [Background] Heimbach D, Luterman A, Burke J, Cram A, Herndon D, Hunt J, Jordan M, McManus W, Solem L, Warden G, et al. Artificial dermis for major burns. A multi-center randomized clinical trial. Ann Surg. 1988 Sep;208(3):313-20. doi: 10.1097/00000658-198809000-00008. PMID 3048216
- [Background] Nguyen DQ, Potokar TS, Price P. An objective long-term evaluation of Integra (a dermal skin substitute) and split thickness skin grafts, in acute burns and reconstructive surgery. Burns. 2010 Feb;36(1):23-8. doi: 10.1016/j.burns.2009.07.011. Epub 2009 Oct 27. PMID 19864070
- [Background] Branski LK, Herndon DN, Pereira C, Mlcak RP, Celis MM, Lee JO, Sanford AP, Norbury WB, Zhang XJ, Jeschke MG. Longitudinal assessment of Integra in primary burn management: a randomized pediatric clinical trial. Crit Care Med. 2007 Nov;35(11):2615-23. doi: 10.1097/01.CCM.0000285991.36698.E2. PMID 17828040
- [Background] Ryan CM, Schoenfeld DA, Malloy M, Schulz JT 3rd, Sheridan RL, Tompkins RG. Use of Integra artificial skin is associated with decreased length of stay for severely injured adult burn survivors. J Burn Care Rehabil. 2002 Sep-Oct;23(5):311-7. doi: 10.1097/00004630-200209000-00002. PMID 12352131
- [Background] Jacoby SM, Bachoura A, Chen NC, Shin EK, Katolik LI. One-stage Integra coverage for fingertip injuries. Hand (N Y). 2013 Sep;8(3):291-5. doi: 10.1007/s11552-013-9513-x. PMID 24426936
- [Background] Burd A, Wong PS. One-stage Integra reconstruction in head and neck defects. J Plast Reconstr Aesthet Surg. 2010 Mar;63(3):404-9. doi: 10.1016/j.bjps.2008.11.105. Epub 2009 Feb 28. PMID 19254877
- [Background] De Angelis B, Gentile P, Tati E, Bottini DJ, Bocchini I, Orlandi F, Pepe G, Di Segni C, Cervelli G, Cervelli V. One-Stage Reconstruction of Scalp after Full-Thickness Oncologic Defects Using a Dermal Regeneration Template (Integra). Biomed Res Int. 2015;2015:698385. doi: 10.1155/2015/698385. Epub 2015 Nov 16. PMID 26649312
- [Background] Demiri E, Papaconstantinou A, Dionyssiou D, Dionyssopoulos A, Kaidoglou K, Efstratiou I. Reconstruction of skin avulsion injuries of the upper extremity with integra((R)) dermal regeneration template and skin grafts in a single-stage procedure. Arch Orthop Trauma Surg. 2013 Nov;133(11):1521-6. doi: 10.1007/s00402-013-1834-2. Epub 2013 Aug 21. PMID 23963344
- [Background] Kosutic D, Beasung E, Dempsey M, Ryan L, Fauzi Z, O'Sullyvan B, Orr D. Single-layer Integra for one-stage reconstruction of scalp defects with exposed bone following full-thickness burn injury: a novel technique. Burns. 2012 Feb;38(1):143-5. doi: 10.1016/j.burns.2011.08.019. Epub 2011 Nov 1. No abstract available. PMID 22047827

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-stage Integra
Started | 2
Completed | 0
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single-stage Integra
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Time to 95% Healing of the Single-stage Reconstructed Skin Graft
Description: 95% healing determined as charted in Standard of Care follow up visits
Time Frame: Up to 12 months
Population: Only two patients were enrolled in this study, and they were withdrawn from the trial prior to initiation of the intervention due to patient characteristics. No data was collected on the two withdrawn patients since the study intervention (graft) was not applied to either subject.
Arm/Group | Single-stage Integra
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency of Complications: Infection, Seroma, Hematoma, Sloughing, and Graft Loss
Description: Compared to the same characteristics of the adjacent (control) 125 cm2 skin graft
Time Frame: Up to 12 months
Population: No patient data was collected due to physician decision to withdraw the patient from the trial prior to initiation of the intervention. No data was collected on the two withdrawn patients since the study intervention (graft) was not applied to either subject.
Arm/Group | Single-stage Integra
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the time of study enrollment (consenting) until the completion of study activities at 12 months (or until the patients were withdrawn from the study).
Arm/Group | Single-stage Integra
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-stage Integra (N=2)
Stroke (Vascular disorders) | 1 (1) — Patient was noted to have left-sided weakness during examination during hospital stay following intervention. Imaging revealed occlusion of the right carotid artery which was consistent with the patient's symptoms

LIMITATIONS AND CAVEATS:
Both subjects were withdrawn by the PI due to their disease state. While subjects were deemed eligible at time of screening and consent upon surgical procedure the patients were deemed too unstable or inappropriate for the study treatment. Patients were notified of this and no further study activities were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03077087/Prot_SAP_000.pdf